CLINICAL TRIAL: NCT01163045
Title: Intraoperative Neuromonitoring and Neurostimulation of the Recurrent Laryngeal Nerve Versus Neurostimulation Alone in Thyroid Surgery: a Randomized Clinical Trial
Brief Title: Intraoperative Neuromonitoring of the Recurrent Laryngeal Nerve Versus Neurostimulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Ottavio Cavicchi, ENT Clinic Policlinico S.Orsola-Malpighi Bologna, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2 - Cavicchi
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-06

CONDITIONS: Thyroidectomy
Keywords: neurostimulation; intraoperative neuromonitoring; recurrent laryngeal nerve; palsy of recurrent laryngeal nerve; RCT
MeSH Terms: interventions — Thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neuromonitoring and neurostimulation (Experimental)
  Interventions: Procedure: thyroidectomy
- neurostimulation of recurrent laryngeal nerve (Experimental)
  Interventions: Procedure: thyroidectomy

INTERVENTIONS:
Procedure: thyroidectomy — total thyroidectomy and lobectomy

SUMMARY:
The purpose of this study is to evaluate if intraoperative neuromonitoring associated to neurostimulation of recurrent laryngeal nerve reduce the rate of recurrent laryngeal palsy respect to neurostimulation alone.

DETAILED DESCRIPTION:
Anatomic and functional preservation of the recurrent laryngeal nerve is a key element of thyroid surgery. Surgical exposure and visual identification of the nerve during thyroid surgery has been shown to provide the best rates of normal postoperative vocal fold function. Nevertheless, identification of the nerve sometimes can be difficult in patients who are heavily scarred or who have undergone previous surgery. Moreover, an anatomical intact nerve does not always correlate with normal vocal fold function. So it is mandatory to identify the nerve and to establish its function. Two techniques are described to facilitate identification of the nerve and to test its function. One is the neurostimulation with laryngeal palpation which is an intermittent monitoring techniques that permits to evaluate the contraction of cricoarytenoid muscle (laryngeal twitch ) after stimulation of RLN or vagal nerve with an electric stimulator probe. More recently some authors have suggested a continuous intraoperative neuromonitoring which provide audio and visual feed back when the nerve is electrically or mechanically stimulated during thyroidectomy. However controversy remains as to whether intraoperative neuromonitoring confers any significant benefit in injury prevention of recurrent laryngeal nerve.

ELIGIBILITY:
Inclusion Criteria:

* Mono or bilateral thyroid surgery

Exclusion Criteria:

* Previous thyroid and parathyroid surgery
* Thyroidectomy with mono or bilateral neck dissection
* Extended thyroidectomy for locally advanced thyroid carcinoma
* Retrosternal goitre
* Minimally invasive thyroid surgery
* Preoperative palsy

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
recurrent laryngeal nerve paralysis

CONTACTS AND LOCATIONS:
Overall Officials: Ottavio O Cavicchi, MD, Study Director — ENT Clinic Ploiclinico S.Orsola-Malpighi Bologna Italy
Locations (1):
- Policlinico S.Orsola-Malpighi ENT Clini University of Bologna Italy, Bologna, Italy/Bologna, Italy

REFERENCES:
- [Result] Barczynski M, Konturek A, Cichon S. Randomized clinical trial of visualization versus neuromonitoring of recurrent laryngeal nerves during thyroidectomy. Br J Surg. 2009 Mar;96(3):240-6. doi: 10.1002/bjs.6417. PMID 19177420
- [Derived] Cavicchi O, Caliceti U, Fernandez IJ, Ceroni AR, Marcantoni A, Sciascia S, Sottili S, Piccin O. Laryngeal neuromonitoring and neurostimulation versus neurostimulation alone in thyroid surgery: a randomized clinical trial. Head Neck. 2012 Feb;34(2):141-5. doi: 10.1002/hed.21681. Epub 2011 Apr 5. PMID 21469244